CLINICAL TRIAL: NCT05452239
Title: Interventional, Randomized, Double-blind, Parallel-group, Placebo-controlled Study of add-on Eptinezumab Treatment to Brief Educational Intervention for the Preventive Treatment of Migraine in Patients With Dual Diagnosis of Migraine and Medication Overuse Headache
Brief Title: A Study of Eptinezumab in Participants With Migraine and Medication Overuse Headache
Acronym: RESOLUTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20007A; 2021-003049-40 (EudraCT Number)
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Results first posted 2025-12-04 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Migraine; Medication Overuse Headache
Keywords: Eptinezumab; Migraine; Medication overuse headache; Brief educational intervention
MeSH Terms: conditions — Migraine Disorders; Headache Disorders, Secondary | interventions — eptinezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eptinezumab (Experimental): Participants will receive an intravenous (IV) infusion of eptinezumab at Week 0 and Week 12.
  Interventions: Drug: Eptinezumab
- Placebo (Placebo Comparator): Participants will receive a single IV infusion of matching placebo to eptinezumab at Week 0. Then, all participants will receive a single IV infusion of eptinezumab at Week 12.
  Interventions: Drug: Eptinezumab; Drug: Placebo

INTERVENTIONS:
Drug: Eptinezumab — Solution for infusion
Drug: Placebo — Solution for infusion
  Arms: Placebo

SUMMARY:
Medication overuse headache (MOH) is a type of headache caused by excessive use of acute headache or migraine medications (medications used to treat a headache or migraine once it begins). Treatment of MOH usually involves reducing the dose of or discontinuing acute medications.

Eptinezumab is a medication used for the preventive treatment of migraine in adults. The main goals of this trial are to learn whether eptinezumab helps reduce the number of days with migraine, the number of days with headache, and acute medication use in adults who have migraine and MOH.

DETAILED DESCRIPTION:
The total study duration from screening visit to safety follow-up visit is approximately 36 weeks and includes a screening period (4 weeks), a placebo-controlled period (12 weeks), an open-label period (12 weeks), and a safety follow-up period (8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of migraine or MOH as defined by IHS ICHD-3 guidelines confirmed at the Screening Visit.
* The participant has ≥8 migraine days per month for each month within the past 3 months prior to the Screening Visit.
* The participant has ≥15 headache days per month for each month within the past 3 months prior to the Screening Visit.
* The participant has had an onset of migraine diagnosis at ≤50 years of age.

Exclusion Criteria:

* The participant has confounding and clinically significant pain syndromes (for example, fibromyalgia, chronic low back pain, and complex regional pain syndrome).
* The participant has a diagnosis of acute or active temporomandibular disorders.
* The participant has a history or diagnosis of chronic tension-type headache, hypnic headache, cluster headache, hemicrania continua, new daily persistent headache, or unusual migraine subtypes such as hemiplegic migraine (sporadic and familial), recurrent painful ophthalmoplegic neuropathy, migraine with brainstem aura, and migraine with neurological accompaniments that are not typical of migraine aura (diplopia, altered consciousness, or long duration).
* The participant has psychosis, bipolar mania, dementia, or any other psychiatric conditions whose symptoms are not controlled or who has not been adequately treated for a minimum of 6 months prior to the Screening Visit.
* The participant has a history of clinically significant cardiovascular disease including uncontrolled hypertension, vascular ischaemia, or thromboembolic events (for example, cerebrovascular accident, deep vein thrombosis, or pulmonary embolism).

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2025-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — HQ_Medinfo@Lundbeck.com
Locations (76):
- United States (6):
  - Clinical Research of Central Florida - ClinEdge - PPDS, Winter Haven, Florida
  - Legacy Clinical Solutions: Tandem Clinical Research LLC - Medical Center - Marrero - ClinEdge - PPDS, Marrero, Louisiana
  - Clinvest - National Ave - Headlands - PPDS, Springfield, Missouri
  - Dent Neurologic Institute - Amherst, Amherst, New York
  - Headache Center - Montefiore Medical Center - BRANY - PPDS, The Bronx, New York
  - Texas Center for Drug Development, Inc, Houston, Texas
- Australia (5):
  - Southern Neurology, Kogarah, New South Wales
  - Mater Adult Hospital, South Brisbane, Queensland
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Health, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Denmark (2):
  - Danish Headache Center, Glostrup Municipality, Capital
  - Sydvestjysk Sygehus Esbjerg, Esbjerg
- France (11):
  - CHU de Nice, Nice, Alpes-Maritimes
  - Assistance Publique Hopitaux de Marseille, Marseille, Bouches-du-Rhône
  - Hôpital Pierre-Paul Riquet, Toulouse, Haute-Garonne
  - Centre Hospitalier Annecy Genevois - Site d'Annecy, Pringy, Haute-Savoie
  - CHRU Nantes, Saint-Herblain, Loire-Atlantique
  - Hôpital Roger Salengro, Lille, Nord
  - Centre Hospitalier Universitaire de Saint Etienne, Saint-Priest-en-Jarez, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Clermont Ferrand -58 Rue Montalembert, Clermont-Ferrand, Puy-de-Dôme
  - Hospices Civils de Lyon - Hôpital Pierre Wertheimer, Bron, Rhône
  - AP-HP - Hopital Lariboisiere, Paris
  - Groupe Hospitalier Paris Saint Joseph, Paris
- Georgia (7):
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center-Gobronidze 10, Tbilisi
  - Ltd Israel-Georgia Medical Research Clinic Helsicore, Tbilisi
  - Pineo Medical Ecosystem, Tbilisi
  - Aversi Clinic LTD, Tbilisi
  - MediClubGeorgia Ltd, Tbilisi
  - S. Khechinashvili University Clinic, Ltd., Tbilisi
  - Multiprofile Clinic Consilium Medulla, Tbilisi
- Germany (8):
  - Klinikverbund Südwest - Kliniken Sindelfingen, Sindelfingen, Baden-Wurttemberg
  - Kopfschmerzzentrum Frankfurt, Frankfurt am Main, Hesse
  - Studienzentrum Nord-West, Westerstede, Lower Saxony
  - Praxis fuer Neurologie, Spezielle Schmerztherapie und Psychotherapie, Essen, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden, Saxony
  - Universitatsklinikum Jena - Am Klinikum 1-Erlanger Allee 101, Jena, Thuringia
  - Universitätsmedizin Greifswald, Greifswald
- Italy (14):
  - ASL 1 Abruzzo - PO Avezzano, Avezzano, Abruzzo
  - Azienda Ospedaliero Universitaria Consorziale Policlinico, Bari, Apulia
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli - Piazza Luigi Miraglia 2, Napoli, Campania
  - IRCCS Istituto delle Scienze Neurologiche - Largo B. Nigrisoli, Bologna, Emilia-Romagna
  - Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Lazio
  - IRCCS San Raffaele, Rome, Lazio
  - Fondazione Policlinico Universitario A Gemelli - Rome - PPDS, Rome, Lazio
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Lombardy
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliera di Perugia - Ospedale Santa Maria della Misericordia, Perugia, Umbria
  - Azienda Ospedaliero Universitaria Di Modena Policlinico, Modena
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone-Palermo-Piazza Delle Cliniche 2, Palermo
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino IRCCS, Pavia
- Leids Universitair Medisch Centrum, Leiden, South Holland, Netherlands
- Norway (4):
  - Akershus Universitetssykehus, Nordbyhagen, Akershus
  - Haukeland Universitetssykehus, Bergen, Hordaland
  - St. Olav's University Hospital, Trondheim, Sør-Trøndelag
  - Oslo Universitetssykehus, Oslo
- Spain (14):
  - Hospital Puerta del Mar, Cadiz, Cádiz
  - C.H. Regional Reina Sofia - PPDS, Córdoba, Córdoba
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario HM Sanchinarro - CIOCC, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Sweden (4):
  - Hallands Sjukhus Halmstad, Halmstad, Halland County
  - Skaneuro Privatmottagning, Lund, Skåne County
  - Karolinska Universitetssjukhuset Huddinge, Huddinge, Stockholm County
  - CTC Clinical Trial Consultants AB, Solna, Stockholm County

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a 12-week placebo-controlled Period followed by a 12-week open-label Period.
Groups:
- Eptinezumab: Participants received an intravenous (IV) infusion of eptinezumab at Baseline (Week 0) during the placebo-controlled period and at Week 12 during the open-label period.
- Placebo: Participants received a single IV infusion of placebo matched to eptinezumab at Week 0 during the placebo-controlled period and an IV infusion of eptinezumab at Week 12 during the open-label period.
Period: Placebo-controlled Period
Arm/Group | Eptinezumab | Placebo
Started | 305 | 303
Received at Least 1 Dose of Study Drug | 303 | 301
Full Analysis Set (FAS) (All randomized participants who received an infusion of the investigational medicinal product (IMP) in the Placebo-controlled Period and had a valid Baseline assessment and at least 1 valid post-Baseline 4-week assessment of monthly migraine days (MMDs) in Weeks 1-12.) | 302 | 300
Completed | 301 | 295
Not Completed | 4 | 8
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Failure to comply with trial procedures | 0 | 1
Not completed — Randomized but not treated | 2 | 2
Not completed — Other than specified | 1 | 1
Period: Open-label Period
Arm/Group | Eptinezumab | Placebo
Started | 300 | 293
Received at Least 1 Dose of Study Drug | 300 | 293
Completed | 294 | 290
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Other than specified | 1 | 2

BASELINE CHARACTERISTICS:
Population: All-Participants-Treated Set (APTS) included all randomized participants who received an infusion of the IMP in the Placebo-controlled Period.
Groups:
- Eptinezumab: Participants received an IV infusion of eptinezumab at Baseline (Week 0) during the placebo-controlled period and at Week 12 during the open-label period.
- Total: Total of all reporting groups
Arm/Group | Eptinezumab | Placebo | Total
Number analyzed (Participants) | 303 | 301 | 604
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (11.95) | 45.2 (12.03) | 45.5 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 264 | 253 | 517
  Male | 39 | 48 | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 151 | 147 | 298
  Race: Black | 3 | 4 | 7
  Race: Asian | 1 | 1 | 2
  Race: Other | 2 | 4 | 6
  Race: Not Collected/Unknown | 146 | 145 | 291
Monthly Migraine Days (MMDs) [Mean (Standard Deviation); unit: days/month] — A Migraine Day was defined as a day with a headache if it belonged to any subgroup of headaches as defined in the outcome measure 1. Population: Full Analysis Set (FAS) included all randomized participants who received an infusion of the IMP in the Placebo-controlled Period and had a valid Baseline assessment and at least 1 valid post-Baseline 4-week assessment of MMDs in Weeks 1-12. Here, MMDs at Baseline are reported.
  days/month
    number analyzed (Participants) | 302 | 300 | 602
    (all) | 21.0 (4.26) | 20.9 (4.28) | 20.9 (4.27)

OUTCOME MEASURES:

1. Primary Outcome: Placebo-controlled Period: Change From Baseline in the Number of MMDs at Weeks 1 - 4
Description: A Migraine Day was defined as a day with a headache if it belonged to any subgroup of headaches that:
  * lasted ≥30 minutes and met following 2 criteria: - ≥2 of following characteristics: unilateral location; pulsating quality, moderate or severe pain intensity, or aggravation by or causing avoidance of routine physical activity; - During headache participant had ≥1 of following: nausea, vomiting, photophobia and phonophobia.
  * lasted ≥30 minutes and participant had an aura with headache.
  * lasted ≥30 minutes and met 2 of following 3 criteria: - lasted 4 hours; - ≥2 of following characteristics: unilateral location; pulsating quality, moderate or severe pain intensity, or aggravation by or causing avoidance of routine physical activity; - During headache participant had ≥1 of following: nausea, vomiting, photophobia and phonophobia.
  * A day with a headache that was successfully treated with a migraine specific treatment.
  * A day with an aura without a headache with medication taken.
Time Frame: Baseline, Weeks 1 - 4
Population: FAS included all randomized participants who received an infusion of the IMP in the Placebo-controlled Period and had a valid Baseline assessment and at least 1 valid post-Baseline 4-week assessment of MMDs in Weeks 1-12. 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: days/month
Groups:
- Placebo-controlled Period: Eptinezumab: Participants received an IV infusion of eptinezumab at Baseline (Week 0) during the placebo-controlled period.
- Placebo-controlled Period: Placebo: Participants received a single IV infusion of placebo matched to eptinezumab at Week 0 during the placebo-controlled period.
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 300 | 299
days/month | -6.85 (0.518) | -3.66 (0.519)
Statistical Analysis 1: Comparison: Placebo-controlled Period: Eptinezumab vs Placebo-controlled Period: Placebo; Analysis was performed using a restricted maximum likelihood (REML)-based mixed model for repeated measurements (MMRM) with Baseline number of MMDs as a continuous covariate and treatment group (eptinezumab versus placebo), month (Weeks 1-4, 5-8, 9-12), country, and previous treatment failures (≤2; >2) as factors. The interaction terms treatment-by-month and previous treatment failures-by-month as well as number of MMDs at baseline-by-month were included; Test type: Other — Testing sequence: 1. Change in MMDs (Weeks 1-4); 2. Change in MMDs (Weeks 1-12); 3. Change in MHDs (Weeks 1-4); 4. Change in MHDs (Weeks 1-12); 5. Participants not fulfilling the ICHD-3 diagnostic criteria for CM nor MOH (Weeks 1-4), 6. Participants not fulfilling the ICHD-3 diagnostic criteria for CM nor MOH (Weeks 1-12), 7. Change in average Daily Pain assessment score (Weeks 1-2); 8. Change in MAMDs (Weeks 1-4), 9. Change in MAMDs (Weeks 1-12); p < 0.0001, Mixed model for repeated measures — Testing continued only if the previous comparison was statistically significant. Threshold for significance: p-value <α, where α = 0.05. Here it is test no. 1 of testing order; Least Square (LS) Mean Difference = -3.20, 95% CI 2-sided [-4.16 to -2.23], Standard Error of Mean 0.490

2. Secondary Outcome: Placebo-controlled Period: Change From Baseline in MMDs at Weeks 1 to 12
Description: as for outcome 1
Time Frame: Baseline, Weeks 1 - 12
Population: FAS included all randomized participants who received an infusion of the IMP in the Placebo-controlled Period and had a valid Baseline assessment and at least 1 valid post-Baseline 4-week assessment of MMDs in Weeks 1-12.
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 302 | 300
days/month | -7.44 (0.508) | -4.50 (0.508)
Statistical Analysis 1: Comparison: Placebo-controlled Period: Eptinezumab vs Placebo-controlled Period: Placebo; Analysis was performed using a REML-based MMRM with Baseline number of MMDs as a continuous covariate and treatment group (eptinezumab versus placebo), month (Weeks 1-4, 5-8, 9-12), country, and previous treatment failures (≤2; >2) as factors. The interaction terms treatment-by-month and previous treatment failures-by-month as well as number of MMDs at baseline-by-month were included; Test type: Other; p < 0.0001, Mixed model for repeated measures — Testing continued only if the previous comparison was statistically significant. Threshold for significance: p-value <α, where α = 0.05. Here it is test no. 2 of testing order; LS Mean Difference = -2.94, 95% CI 2-sided [-3.86 to -2.02], Standard Error of Mean 0.469

3. Secondary Outcome: Placebo-controlled Period: Change From Baseline in the Number of Monthly Headache Days (MHDs) at Weeks 1 to 4 and Weeks 1 to 12
Description: A headache day was defined as a day with a headache that lasted ≥30 minutes or that met the definition of a migraine day (as defined in outcome measure 1).
Time Frame: Baseline, Weeks 1 - 4 and Weeks 1 - 12
Population: FAS included all randomized participants who received an infusion of the IMP in the Placebo-controlled Period and had a valid Baseline assessment and at least 1 valid post-Baseline 4-week assessment of MMDs in Weeks 1-12. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 302 | 300
days/month
  Change at Weeks 1-4: number analyzed (Participants) | 300 | 299
  Change at Weeks 1-4 | -6.54 (0.502) | -3.40 (0.502)
  Change at Weeks 1-12 | -7.38 (0.497) | -4.45 (0.497)
Statistical Analysis 1: Comparison: Placebo-controlled Period: Eptinezumab vs Placebo-controlled Period: Placebo; Analysis was performed using a REML-based MMRM with Baseline number of MHDs as a continuous covariate and treatment group (eptinezumab versus placebo), month (Weeks 1-4, 5-8, 9-12), country, and previous treatment failures (≤2; >2) as factors. The interaction terms treatment-by-month and previous treatment failures-by-month as well as number of MHDs at baseline-by-month were included; Test type: Other; p < 0.0001, Mixed model for repeated measures — Testing continued only if the previous comparison was statistically significant. Threshold for significance: p-value <α, where α = 0.05. Here it is test no. 3 of testing order; LS Mean Difference = -3.15, 95% CI 2-sided [-4.07 to -2.22], Standard Error of Mean 0.471 — Change From Baseline in the Number of MHDs at Weeks 1 to 4: Eptinezumab vs. Placebo
Statistical Analysis 2: Comparison: Placebo-controlled Period: Eptinezumab vs Placebo-controlled Period: Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Other; p < 0.0001, Mixed model for repeated measures — Testing continued only if the previous comparison was statistically significant. Threshold for significance: p-value <α, where α = 0.05. Here it is test no. 4 of testing order; LS Mean Difference = -2.93, 95% CI 2-sided [-3.83 to -2.02], Standard Error of Mean 0.460 — Change From Baseline in the Number of MHDs at Weeks 1 to 12 (averaged over three 4-week intervals): Eptinezumab vs. Placebo

4. Secondary Outcome: Placebo-controlled Period: Percentage of Participants Not Fulfilling the International Classification of Headache Disorders, 3rd Edition (ICHD-3) Diagnostic Criteria for Chronic Migraine (CM) Nor Medication Overuse Headache (MOH)
Description: CM: - Headache on ≥15 days/month for >3 months. - Participants had experienced ≥5 attacks that fulfilled the criteria for either migraine without aura or with aura. - On ≥8 days/month for >3 months, headache meeting the criteria for either: Migraine without aura (headache with ≥2 of these features: unilateral location, pulsating quality, moderate to severe pain, or aggravation by physical activity; plus either nausea/vomiting or photophobia/phonophobia); Migraine with aura (headache preceded or accompanied by transient focal neurological symptoms, such as visual or sensory disturbances); or headache believed to be migraine by participant and relieved by a triptan or ergot derivative. - Not better accounted for by another ICHD-3 diagnosis.
  MOH: Headache occurring on ≥15 days/month with a pre-existing headache. - Regular overuse for >3 months of ≥1 drug that can be taken for acute and/or symptomatic treatment of headache. - Not better accounted for by another ICHD-3 diagnosis.
Time Frame: Weeks 1 - 4 and Weeks 1 - 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 302 | 300
percentage of participants
  Weeks 1-4: number analyzed (Participants) | 299 | 298
  Weeks 1-4 | 37.8 | 18.1
  Weeks 1-12 | 27.2 | 12.7
Statistical Analysis 1: Comparison: Placebo-controlled Period: Eptinezumab vs Placebo-controlled Period: Placebo; The logistic regression model with baseline MMDs as a covariate, and treatment group (eptinezumab versus placebo), country and previous treatment failures (≤2, >2) as categorical variables based on the eDiary data collected over Weeks 1-4, Weeks 5-8, Weeks 9-12 and over Weeks 1-12 separately, was fitted using the maximum likelihood method and the logit link function; Test type: Other; p < 0.0001, Regression, Logistic — Testing continued only if the previous comparison was statistically significant. Threshold for significance: p-value <α, where α = 0.05. Here it is test no. 5 of testing order; Odds Ratio (OR) = 3.26, 95% CI 2-sided [2.18 to 4.94] — Percentage of participants not fulfilling the ICHD-3 Diagnostic Criteria for CM nor MOH at Weeks 1 to 4: Eptinezumab vs. Placebo
Statistical Analysis 2: Comparison: Placebo-controlled Period: Eptinezumab vs Placebo-controlled Period: Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Other; p < 0.0001, Regression, Logistic — Testing continued only if the previous comparison was statistically significant. Threshold for significance: p-value <α, where α = 0.05. Here it is test no. 6 of testing order; Odds Ratio (OR) = 3.05, 95% CI 2-sided [1.93 to 4.90] — Percentage of participants not fulfilling the ICHD-3 Diagnostic Criteria for CM nor MOH at Weeks 1 - 12 (averaged over three 4-week intervals): Eptinezumab vs. Placebo

5. Secondary Outcome: Placebo-controlled Period: Change From Baseline in Average Daily Pain Assessment Score at Weeks 1 to 2
Description: Daily Pain assessment data were collected in the headache electronic diary (eDiary) via the question "What was the worst pain intensity of this headache today?". The pain intensity assessment was collected on a 3-point scale: Mild (score = 1), Moderate (score = 2), and Severe (score = 3). For each day, the Daily Pain assessment score was derived by averaging the worst pain intensity over all headaches of that day. For days on which no headaches took place during the relevant period, the Daily Pain score was given as a score of 0. The average Daily Pain score was calculated using the Daily Pain assessments collected during Weeks 1-2.
Time Frame: Baseline, Weeks 1 - 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 302 | 300
units on a scale | -0.58 (0.048) | -0.27 (0.048)
Statistical Analysis 1: Comparison: Placebo-controlled Period: Eptinezumab vs Placebo-controlled Period: Placebo; Analysis of covariance (ANCOVA) was performed with the average Daily Pain at baseline as a covariate and including treatment group, country, and previous treatment failures, as categorical variables; Test type: Other; p < 0.0001, ANCOVA — Testing continued only if the previous comparison was statistically significant. Threshold for significance: p-value <α, where α = 0.05. Here it is test no. 7 of testing order; LS Mean Difference = -0.31, 95% CI 2-sided [-0.39 to -0.22], Standard Error of Mean 0.044

6. Secondary Outcome: Placebo-controlled Period: Change From Baseline in Monthly Days With Acute Migraine Medication Use at Weeks 1 to 4 and Weeks 1 to 12
Description: Acute migraine medication included those medications classified as opioid, barbiturates, ergotamine, triptan, non-opioid analgesic, and combination of analgesic ingredients.
Time Frame: Baseline, Weeks 1 - 4 and Weeks 1 - 12
Population: FAS included all randomized participants who received an infusion of the IMP in the Placebo-controlled Period and had a valid Baseline assessment and at least 1 valid post-Baseline 4-week assessment of MMDs in Weeks 1-12. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 302 | 300
days/month
  Change at Weeks 1-4: number analyzed (Participants) | 299 | 298
  Change at Weeks 1-4 | -11.32 (0.508) | -7.69 (0.509)
  Change at Weeks 1-12 | -11.18 (0.490) | -7.83 (0.490)
Statistical Analysis 1: Comparison: Placebo-controlled Period: Eptinezumab vs Placebo-controlled Period: Placebo; Analysis was performed using a REML-based MMRM with Baseline number of monthly days with acute migraine medication use as a continuous covariate and treatment group (eptinezumab versus placebo), month (Weeks 1-4, 5-8, 9-12), country, and previous treatment failures (≤2; >2) as factors. The interaction terms treatment-by-month and previous treatment failures-by-month as well as number of monthly days with acute migraine medication use at baseline-by-month were included; Test type: Other; p < 0.0001, Mixed model for repeated measures — Testing continued only if the previous comparison was statistically significant. Threshold for significance: p-value <α, where α = 0.05. Here it is test no. 8 of testing order; LS Mean Difference = -3.63, 95% CI 2-sided [-4.59 to -2.67], Standard Error of Mean 0.487 — Change from baseline in monthly days with acute migraine medication use at Weeks 1 to 4: Eptinezumab vs. Placebo
Statistical Analysis 2: Comparison: Placebo-controlled Period: Eptinezumab vs Placebo-controlled Period: Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Other; p < 0.0001, Mixed model for repeated measures — Testing continued only if the previous comparison was statistically significant. Threshold for significance: p-value <α, where α = 0.05. Here it is test no. 9 of testing order; LS Mean Difference = -3.35, 95% CI 2-sided [-4.23 to -2.48], Standard Error of Mean 0.447 — Change from baseline in monthly days with acute migraine medication use at Weeks 1 - 12 (averaged over three 4-week intervals): Eptinezumab vs. Placebo

7. Secondary Outcome: Open-label Period: Change From Baseline in MMDs at Weeks 13-16, 17-20, and 21-24
Description: as for outcome 1
Time Frame: Baseline, Weeks 13-16, 17-20, and 21-24
Population: All-Participants-Treated-Open-Label Set (APTS-OL) included all randomized participants who received an infusion of the IMP in the Open-label Period. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: days/month
Groups:
- Open-label Period: Eptinezumab - Eptinezumab: Participants who received eptinezumab during the placebo-controlled period, received an IV infusion of eptinezumab at Week 12 during the open-label period.
- Open-label Period: Placebo - Eptinezumab: Participants who received placebo during the placebo-controlled period, received an IV infusion of eptinezumab at Week 12 during the open-label period.
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 293 | 285
days/month
  Change at Weeks 13-16 | -10.23 (7.167) | -10.08 (7.136)
  Change at Weeks 17-20: number analyzed (Participants) | 286 | 281
  Change at Weeks 17-20 | -10.29 (7.093) | -10.29 (7.301)
  Change at Weeks 21-24: number analyzed (Participants) | 277 | 278
  Change at Weeks 21-24 | -9.24 (7.220) | -9.30 (7.602)

8. Secondary Outcome: Open-label Period: Change From Baseline in the Number of MHDs at Weeks 13-16, 17-20, and 21-24
Description: as for outcome 3
Time Frame: Baseline, at Weeks 13-16, 17-20, and 21-24
Population: APTS-OL included all randomized participants who received an infusion of the IMP in the Open-label Period. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: days/month
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 293 | 285
days/month
  Change at Weeks 13-16 | -10.31 (7.113) | -9.99 (7.082)
  Change at Weeks 17-20: number analyzed (Participants) | 286 | 281
  Change at Weeks 17-20 | -10.46 (6.941) | -10.34 (7.253)
  Change at Weeks 21-24: number analyzed (Participants) | 277 | 278
  Change at Weeks 21-24 | -9.46 (7.206) | -9.47 (7.382)

9. Secondary Outcome: Open-label Period: Percentage of Participants Not Fulfilling the ICHD-3 Diagnostic Criteria for CM Nor MOH at Weeks 13 to 24
Description: as for outcome 4
Time Frame: Weeks 13 - 24
Population: APTS-OL included all randomized participants who received an infusion of the IMP in the Open-label Period. 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 296 | 291
percentage of participants | 38.9 | 40.2

10. Secondary Outcome: Open-label Period: Change From Baseline in Average Daily Pain Assessment Score at Weeks 13-16, 17-20, and 21-24
Description: Daily Pain assessment data were collected in the headache eDiary via the question "What was the worst pain intensity of this headache today?". The pain intensity assessment was collected on a 3-point scale: Mild (score = 1), Moderate (score = 2), and Severe (score = 3). For each day, the Daily Pain assessment score was derived by averaging the worst pain intensity over all headaches of that day. For days on which no headaches took place during the relevant period, the Daily Pain score was given as a score of 0. The average Daily Pain score was calculated using the Daily Pain assessments collected during Weeks 13-16, 17-20, and 21-24.
Time Frame: Baseline, Weeks 13-16, 17-20, and 21-24
Population: APTS-OL included all randomized participants who received an infusion of the IMP in the Open-label Period. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 300 | 293
units on a scale
  Change at Weeks 13-16 | -0.90 (0.628) | -0.90 (0.602)
  Change at Weeks 17-20: number analyzed (Participants) | 296 | 289
  Change at Weeks 17-20 | -0.88 (0.641) | -0.89 (0.630)
  Change at Weeks 21-24: number analyzed (Participants) | 292 | 286
  Change at Weeks 21-24 | -0.84 (0.638) | -0.81 (0.667)

11. Secondary Outcome: Open-label Period: Change From Baseline in Monthly Days With Acute Migraine Medication Use at Weeks 13-16, 17-20, and 21-24
Description: Acute migraine medication included paracetamol, triptans, ergotamine, combination of non-opioid analgesics, individual non-opioid analgesics, and nonsteroidal anti-inflammatory drugs (NSAIDs). Barbiturates and/or opioid analgesics were allowed when considered medically indicated providing its use does not exceed 4 days per month.
Time Frame: Baseline, Weeks 13-16, 17-20, and 21-24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days/month
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 289 | 282
days/month
  Change at Weeks 13-16 | -12.08 (6.738) | -11.67 (6.470)
  Change at Weeks 17-20: number analyzed (Participants) | 285 | 280
  Change at Weeks 17-20 | -11.82 (6.690) | -11.39 (7.080)
  Change at Weeks 21-24: number analyzed (Participants) | 275 | 273
  Change at Weeks 21-24 | -10.96 (6.693) | -10.44 (7.338)

12. Secondary Outcome: Placebo-controlled Period: Percentage of Participants Not Fulfilling the ICHD-3 Diagnostic Criteria for CM at Weeks 1 to 4 and Weeks 1 to 12
Description: CM: - Headache on ≥15 days/month for >3 months. - Participants had experienced ≥5 attacks that fulfilled the criteria for either migraine without aura or with aura. - On ≥8 days/month for >3 months, headache meeting the criteria for either: Migraine without aura (headache with ≥2 of these features: unilateral location, pulsating quality, moderate to severe pain, or aggravation by physical activity; plus either nausea/vomiting or photophobia/phonophobia); Migraine with aura (headache preceded or accompanied by transient focal neurological symptoms, such as visual or sensory disturbances); or headache believed to be migraine by participant and relieved by a triptan or ergot derivative. - Not better accounted for by another ICHD-3 diagnosis.
Time Frame: Weeks 1 - 4 and Weeks 1 - 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 302 | 300
percentage of participants
  Weeks 1-4: number analyzed (Participants) | 300 | 299
  Weeks 1-4 | 55.0 | 32.4
  Weeks 1-12 | 44.4 | 23.0

13. Secondary Outcome: Placebo-controlled Period: Percentage of Participants Not Fulfilling the ICHD-3 Diagnostic Criteria for MOH at Weeks 1 to 4 and Weeks 1 to 12
Description: MOH: Headache occurring on ≥15 days/month with a pre-existing headache. - Regular overuse for >3 months of ≥1 drug that can be taken for acute and/or symptomatic treatment of headache. - Not better accounted for by another ICHD-3 diagnosis.
Time Frame: Weeks 1 - 4 and Weeks 1 - 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 302 | 300
percentage of participants
  Weeks 1-4: number analyzed (Participants) | 299 | 298
  Weeks 1-4 | 52.2 | 31.9
  Weeks 1-12 | 40.1 | 24.0

14. Secondary Outcome: Placebo-controlled Period: Change From Baseline in MMDs With Use of Acute Headache Medication at Weeks 1 to 12
Description: as for outcome 1
Time Frame: Baseline, Weeks 1 - 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 302 | 300
days/month | -10.32 (0.481) | -7.16 (0.481)

15. Secondary Outcome: Placebo-controlled Period: Change From Baseline in Monthly Days With Triptan or Ergotamine Medication Use at Weeks 1 to 12
Time Frame: Baseline, Weeks 1 - 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 302 | 300
days/month | -8.35 (0.411) | -5.49 (0.409)

16. Secondary Outcome: Open-label Period: Change From Baseline in Monthly Days With Triptan or Ergotamine Medication Use at Weeks 13-16, 17-20, and 21-24
Time Frame: Baseline, Weeks 13-16, 17-20, and 21-24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days/month
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 289 | 282
days/month
  Change at Weeks 13-16 | -8.70 (6.736) | -8.79 (6.781)
  Change at Weeks 17-20: number analyzed (Participants) | 285 | 280
  Change at Weeks 17-20 | -8.24 (6.540) | -8.31 (6.982)
  Change at Weeks 21-24: number analyzed (Participants) | 275 | 273
  Change at Weeks 21-24 | -7.43 (6.505) | -7.56 (6.700)

17. Secondary Outcome: Placebo-controlled Period: Change From Baseline in Monthly Days With Individual Non-opioid Analgesics or Non-steroidal Anti-inflammatory Drug (NSAID) Medication Use at Weeks 1 to 12
Time Frame: Baseline, Weeks 1 - 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 294 | 295
days/month | -5.94 (0.402) | -4.80 (0.402)

18. Secondary Outcome: Open-label Period: Change From Baseline in Monthly Days With Individual Non-opioid Analgesics or NSAID Medication Use at Weeks 13-16, 17-20, and 21-24
Time Frame: Baseline, Weeks 13-16, 17-20, and 21-24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days/month
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 289 | 282
days/month
  Change at Weeks 13-16 | -6.55 (7.205) | -6.66 (7.108)
  Change at Weeks 17-20: number analyzed (Participants) | 285 | 280
  Change at Weeks 17-20 | -6.65 (7.193) | -6.62 (7.316)
  Change at Weeks 21-24: number analyzed (Participants) | 275 | 273
  Change at Weeks 21-24 | -6.18 (7.018) | -6.44 (7.468)

19. Secondary Outcome: Placebo-controlled Period: Change From Baseline in Monthly Days With Combination Non-opioid Analgesics Medication Use at Weeks 1 to 12
Time Frame: Baseline, Weeks 1 - 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 294 | 295
days/month | -1.24 (0.202) | -1.12 (0.201)

20. Secondary Outcome: Placebo-controlled Period: Number of Participants With Migraine on the Day After Dosing
Time Frame: Day 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 302 | 300
Participants | 162 | 203

21. Secondary Outcome: Placebo-controlled Period: Percentage of Participants With ≥50% Reduction From Baseline in MMDs at Weeks 1 to 4 and Weeks 1 to 12
Description: as for outcome 1
Time Frame: Baseline to Weeks 1 - 4 and 1 - 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 302 | 300
percentage of participants
  Weeks 1-4: number analyzed (Participants) | 300 | 299
  Weeks 1-4 | 36.7 | 13.7
  Weeks 1-12 | 40.4 | 18.0

22. Secondary Outcome: Placebo-controlled Period: Percentage of Participants With ≥75% Reduction From Baseline in MMDs at Weeks 1 to 4 and Weeks 1 to 12
Description: as for outcome 1
Time Frame: Baseline to Weeks 1 - 4 and 1 - 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 302 | 300
percentage of participants
  Weeks 1-4: number analyzed (Participants) | 300 | 299
  Weeks 1-4 | 13.0 | 4.3
  Weeks 1-12 | 12.9 | 5.3

23. Secondary Outcome: Placebo-controlled Period: Percentage of Participants With ≥50% Reduction From Baseline in MHDs at Weeks 1 to 4 and Weeks 1 to 12
Description: as for outcome 3
Time Frame: Baseline to Weeks 1 - 4 and 1 - 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 302 | 300
percentage of participants
  Weeks 1-4: number analyzed (Participants) | 300 | 299
  Weeks 1-4 | 33.0 | 11.0
  Weeks 1-12 | 35.8 | 15.3

24. Secondary Outcome: Placebo-controlled Period: Percentage of Participants With ≥75% Reduction From Baseline in MHDs at Weeks 1 to 4 and Weeks 1 to 12
Description: as for outcome 3
Time Frame: Baseline to Weeks 1 - 4 and 1 - 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 302 | 300
percentage of participants
  Weeks 1-4: number analyzed (Participants) | 300 | 299
  Weeks 1-4 | 9.3 | 3.3
  Weeks 1-12 | 10.9 | 5.3

25. Secondary Outcome: Placebo-controlled Period: Change From Baseline in Percentage of Migraine Attacks With Severe Pain Intensity at Weeks 1 to 4 and Weeks 1 to 12
Description: A migraine that fulfilled the criteria for a migraine, was referred to as a migraine attack.
Time Frame: Baseline to Weeks 1 - 4 and 1 - 12
Population: FAS included all randomized participants who received an infusion of the IMP in the Placebo-controlled Period and had a valid Baseline assessment and at least 1 valid post-Baseline 4-week assessment of MMDs in Weeks 1-12. 'Overall number of participants analyzed' = participants analyzed for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: percentage of migraine attacks
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 299 | 297
percentage of migraine attacks
  Change at Weeks 1-4 | -10.30 (1.912) | -1.60 (1.916)
  Change at Weeks 1-12: number analyzed (Participants) | 289 | 288
  Change at Weeks 1-12 | -5.21 (1.859) | -1.60 (1.860)

26. Secondary Outcome: Placebo-controlled Period: Change From Baseline in Percentages of Headache Episodes With Severe Pain Intensity at Weeks 1 to 4 and Weeks 1 to 12
Description: A non-migraine headache that lasted ≥30 minutes or a migraine headache, was referred to as a headache episode.
Time Frame: Baseline to Weeks 1 - 4 and 1 - 12
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: percentage of headache episodes
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 300 | 297
percentage of headache episodes
  Change at Weeks 1-4 | -11.78 (1.867) | -3.36 (1.872)
  Change at Weeks 1-12: number analyzed (Participants) | 291 | 289
  Change at Weeks 1-12 | -6.99 (1.822) | -2.79 (1.825)

27. Secondary Outcome: Placebo-controlled Period: Patient Global Impression of Change (PGIC) Score at Weeks 4 and 12
Description: The PGIC is a single, participant-reported item reflecting the participant's impression of change in his/her disease status since the start of the study (that is, in relation to activity limitations, symptoms, emotions, and overall quality of life). Participants rated their impression of change in disease status on a 7-point scale (1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse) where a higher score indicated worsening. Score ranges from 1 (Very Much Improved) to 7 (Very Much Worse). Lower scores indicate better health status.
Time Frame: Weeks 4 and 12
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 288 | 284
units on a scale
  Week 4: number analyzed (Participants) | 279 | 274
  Week 4 | 2.62 (0.100) | 3.63 (0.100)
  Week 12 | 2.64 (0.101) | 3.54 (0.101)

28. Secondary Outcome: Open-label Period: PGIC Score at Week 24
Description: as for outcome 27
Time Frame: Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 283 | 277
units on a scale | 2.3 (1.18) | 2.3 (1.20)

29. Secondary Outcome: Placebo-controlled Period: Most Bothersome Symptom (MBS) Score at Week 12
Description: Participants were asked about their most bothersome symptom associated with their migraines during the Baseline Visit. Participants were asked to rate the improvement in this symptom from baseline on a 7-point scale (1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse) where a high score indicated worsening. Score ranges from 1 (Very Much Improved) to 7 (Very Much Worse). Lower scores indicate better health status. The MBS areas included: nausea, vomiting, sensitivity to light, sensitivity to sound, mental cloudiness, fatigue, pain with activity, mood changes, and other symptoms.
Time Frame: Week 12
Population: FAS included all randomized participants who received an infusion of the IMP in the Placebo-controlled Period and had a valid Baseline assessment and at least 1 valid post-Baseline 4-week assessment of MMDs in Weeks 1-12. 'Overall number of participants analyzed' = participants analyzed for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 288 | 283
units on a scale | 2.87 (0.106) | 3.59 (0.107)

30. Secondary Outcome: Open-label Period: MBS Score at Week 24
Description: as for outcome 29
Time Frame: Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 283 | 277
units on a scale | 2.6 (1.22) | 2.6 (1.25)

31. Secondary Outcome: Placebo-controlled Period: Change From Baseline in Headache Impact Test (HIT-6) Total Score at Weeks 4 and 12
Description: The HIT-6 (version 1.0) is a Likert-type, self-reporting questionnaire designed to assess the impact of an occurring headache and its effect on the ability to function normally in daily life. The HIT-6 contains 6 questions, each item was rated from never to always with the following response scores: never = 6, rarely = 8, sometimes = 10, very often = 11, and always = 13. The total score for the HIT-6 was the sum of each response score ranging from 36 to 78. The life impact derived from the total score was described as followed: severe (≥60), substantial (56-59), some (50-55), little to none (≤49).
Time Frame: Baseline, Weeks 4 and 12
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 279 | 274
units on a scale
  Change at Week 4: number analyzed (Participants) | 276 | 268
  Change at Week 4 | -6.5 (7.25) | -2.6 (5.30)
  Change at Week 12 | -7.4 (8.60) | -3.9 (6.42)

32. Secondary Outcome: Open-label Period: Change From Baseline in HIT-6 Total Score at Week 24
Description: as for outcome 31
Time Frame: Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 274 | 265
units on a scale | -8.1 (8.21) | -7.6 (7.74)

33. Secondary Outcome: Placebo-controlled Period: Change From Baseline in Modified Migraine Disability Assessment (mMIDAS) Total Score at Weeks 4 and 12
Description: The mMIDAS is a self-administered questionnaire that contains 7 questions about the headache a participant had in the previous month. The first 5 questions assess the impact of migraine on 3 domains of daily activity: 2 questions for paid work or schoolwork, 2 questions for household work, and 1 question for family, social and leisure activities. The 2 questions for each of the first two groups assess, respectively, the number of days off due to headache, and the number of days in which the productivity was reduced by half or more. mMIDAS total score was derived from the sum of the answers on the first 5 questions. Total score ranged from 0 (little/no disability) to 20 (severe disability) with higher scores indicating more severe disability.
Time Frame: Baseline, Weeks 4 and 12
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 276 | 271
units on a scale
  Change at Week 4: number analyzed (Participants) | 274 | 263
  Change at Week 4 | -14.73 (1.475) | -6.62 (1.476)
  Change at Week 12 | -13.83 (1.494) | -8.76 (1.496)

34. Secondary Outcome: Open-label Period: Change From Baseline in mMIDAS Total Score at Week 24
Description: as for outcome 33
Time Frame: Baseline, Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 270 | 263
units on a scale | -17.3 (20.71) | -15.2 (19.69)

35. Secondary Outcome: Placebo-controlled Period: Change From Baseline in Migraine-Specific Quality of Life Questionnaire, Version 2.1 (MSQ v2.1) Subscores (Role Function-Restrictive, Role Function-Preventive, Emotional Function) at Weeks 4 and 12
Description: The MSQ v2.1 is a participant-reported outcome designed to assess the quality of life in participants with migraine. It consists of 14 items covering 3 domains: role function restrictive (7 items); role function preventive (4 items); and emotional function (3 items). Each item was scored on a 6-point scale ranging from 1 (none of the time) to 6 (all of the time). Raw domain scores were summed and transformed to a 0-to-100-point scale. Higher scores indicated better quality of life.
Time Frame: Baseline, Weeks 4 and 12
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 276 | 267
units on a scale
  Change at Week 4: Role function- restrictive: number analyzed (Participants) | 272 | 256
  Change at Week 4: Role function- restrictive | 24.04 (1.898) | 10.15 (1.902)
  Change at Week 12: Role function- restrictive | 22.55 (1.873) | 11.79 (1.877)
  Change at Week 4: Role function- preventive: number analyzed (Participants) | 272 | 256
  Change at Week 4: Role function- preventive | 18.58 (1.862) | 7.88 (1.864)
  Change at Week 12: Role function- preventive | 17.96 (1.834) | 10.16 (1.836)
  Change at Week 4: Emotional function: number analyzed (Participants) | 272 | 256
  Change at Week 4: Emotional function | 23.82 (2.143) | 10.11 (2.145)
  Change at Week 12: Emotional function | 22.06 (2.188) | 11.67 (2.193)

36. Secondary Outcome: Open-label Period: Change From Baseline in MSQ v2.1 Subscores (Role Function-Restrictive, Role Function-Preventive, Emotional Function) at Week 24
Description: as for outcome 35
Time Frame: Baseline, Weeks 24
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 270 | 257
units on a scale
  Role function- restrictive | 26.38 (23.302) | 26.33 (24.159)
  Role function- preventive | 20.6 (23.61) | 20.7 (22.85)
  Emotional function | 26.86 (27.806) | 26.54 (28.385)

37. Secondary Outcome: Placebo-controlled Period: Change From Baseline in Euroqol 5 Dimension - 5 Levels (EQ-5D-5L) Visual Analogue Scale (VAS) Score at Weeks 4 and 12
Description: The EQ-5D-5L VAS measures participant's self-rated health-related quality of life on a VAS. The VAS score ranged from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline, Weeks 4 and 12
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 276 | 264
units on a scale
  Change at Week 4: number analyzed (Participants) | 270 | 252
  Change at Week 4 | 5.09 (1.561) | 0.49 (1.574)
  Change at Week 12 | 7.43 (1.526) | 2.23 (1.540)

38. Secondary Outcome: Open-label Period: Change From Baseline in EQ-5D-5L VAS Score at Week 24
Description: as for outcome 37
Time Frame: Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 268 | 256
units on a scale | 5.9 (22.69) | 3.9 (22.10)

39. Secondary Outcome: Placebo-controlled Period: Change From Baseline in Work Productivity and Activity Impairment: Migraine (WPAI:M) Sub-scores (Absenteeism, Presenteeism, Work Productivity Loss, Activity Impairment) at Week 12
Description: The WPAI Questionnaire is a participant-reported instrument developed to measure the impact on work productivity and regular activities attributable to a specific health problem (migraine). Recall period is the past 7 days. It contains 6 items that measure: 1) employment status, 2) hours missed from work due to the specific health problem, 3) hours missed from work for other reasons, 4) hours actually worked, 5) degree health affected productivity while working, and 6) degree health affected productivity in regular unpaid activities. Four scores were calculated from the responses to these 6 items: absenteeism, presenteeism, work productivity loss, and activity impairment. Scores were calculated as impairment percentages (0-100%), with higher numbers indicating greater impairment and less productivity, that is, worse outcomes.
Time Frame: Baseline, Week 12
Population: FAS included all randomized participants who received an infusion of the IMP in the Placebo-controlled Period and had a valid Baseline assessment and at least 1 valid post-Baseline 4-week assessment of MMDs in Weeks 1-12. 'Overall number of participants analyzed' = participants analyzed for this outcome measure. 'Number analyzed' = participants evaluable at specified category.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 276 | 263
units on a scale
  Absenteeism: number analyzed (Participants) | 169 | 162
  Absenteeism | -4.73 (2.342) | -1.18 (2.324)
  Presenteeism: number analyzed (Participants) | 154 | 156
  Presenteeism | -19.10 (2.602) | -10.12 (2.544)
  Work productivity loss: number analyzed (Participants) | 154 | 156
  Work productivity loss | -19.88 (2.790) | -9.04 (2.727)
  Activity impairment | -18.87 (2.065) | -10.42 (2.079)

40. Secondary Outcome: Open-label Period: Change From Baseline in WPAI:M Sub-scores (Absenteeism, Presenteeism, Work Productivity Loss, Activity Impairment) at Week 24
Description: as for outcome 39
Time Frame: Baseline, Week 24
Population: APTS-OL included all randomized participants who received an infusion of the IMP in the Open-label Period. 'Overall number of participants analyzed' = participants analyzed for this outcome measure. 'Number analyzed' = participants evaluable at specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 268 | 256
units on a scale
  Absenteeism: number analyzed (Participants) | 161 | 145
  Absenteeism | -9.22 (27.236) | -4.75 (25.007)
  Presenteeism: number analyzed (Participants) | 152 | 136
  Presenteeism | -18.8 (28.41) | -22.7 (27.58)
  Work productivity loss: number analyzed (Participants) | 152 | 136
  Work productivity loss | -20.54 (29.162) | -24.18 (29.102)
  Activity impairment | -19.6 (28.14) | -21.0 (28.73)

41. Secondary Outcome: Placebo-controlled Period: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Subscale (Depression and Anxiety) Scores at Weeks 4 and 12
Description: The HADS is a participant-rated scale designed to assess psychological distress in non-psychiatric participants. The HADS consists of 2 sub-scales: depression and anxiety. Each sub-scale contains 7 items, and each item was rated from 0 (absent) to 3 (maximum severity). The total score of each sub-scale ranged from 0 (absent) to 21 (maximum severity). Higher scores indicated higher severity.
Time Frame: Baseline, Weeks 4 and 12
Population: as for outcome 39
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 276 | 264
units on a scale
  Change at Week 4: Total Depression Score: number analyzed (Participants) | 272 | 252
  Change at Week 4: Total Depression Score | -1.59 (0.294) | -0.61 (0.296)
  Change at Week 12: Total Depression Score | -1.82 (0.300) | -0.64 (0.302)
  Change at Week 4: Total Anxiety Score: number analyzed (Participants) | 272 | 252
  Change at Week 4: Total Anxiety Score | -1.32 (0.262) | -0.49 (0.263)
  Change at Week 12: Total Anxiety Score | -1.37 (0.257) | -0.40 (0.257)

42. Secondary Outcome: Open-label Period: Change From Baseline in HADS Subscale (Depression and Anxiety) Scores at Week 24
Description: as for outcome 41
Time Frame: Baseline, Week 24
Population: APTS-OL included all randomized participants who received an infusion of the IMP in the Open-label Period. 'Overall number of participants analyzed' = participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 269 | 256
units on a scale
  Total Depression Score | -2.1 (3.78) | -1.3 (3.88)
  Total Anxiety Score | -2.0 (3.36) | -1.1 (3.54)

43. Secondary Outcome: Placebo-controlled Period: Treatment Satisfaction Questionnaire for Medicine - 9 Items (TSQM-9) Score at Weeks 4 and 12
Description: TSQM is a 14-item instrument consisting of four scales: effectiveness scale (questions 1 to 3), side effects scale (questions 4 to 8), convenience scale (questions 9 to 11) and global satisfaction scale (questions 12 to 14). In TSQM-9, the five items related to side effects of medication were not included. The scores were computed by adding items for each domain. The lowest possible score was subtracted from this composite score and divided by the greatest possible score minus the lowest possible score. This provided a transformed score between 0 and 1 that was then multiplied by 100. TSQM-9 domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domain.
Time Frame: Weeks 4 and 12
Population: as for outcome 39
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 288 | 281
units on a scale
  Week 4: Effectiveness Score: number analyzed (Participants) | 275 | 267
  Week 4: Effectiveness Score | 58.21 (2.228) | 39.01 (2.236)
  Week 12: Effectiveness Score | 57.95 (2.264) | 40.89 (2.278)
  Week 4: Convenience Score: number analyzed (Participants) | 275 | 267
  Week 4: Convenience Score | 69.60 (1.736) | 63.62 (1.743)
  Week 12: Convenience Score | 69.42 (1.786) | 63.12 (1.797)
  Week 4: Overall Satisfaction Score: number analyzed (Participants) | 275 | 267
  Week 4: Overall Satisfaction Score | 59.56 (2.094) | 43.57 (2.099)
  Week 12: Overall Satisfaction Score | 62.54 (2.136) | 46.98 (2.146)

44. Secondary Outcome: Open-label Period: TSQM-9 Score at Week 24
Description: as for outcome 43
Time Frame: Baseline, Week 24
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 281 | 276
units on a scale
  Effectiveness Score | 63.23 (28.684) | 62.50 (27.896)
  Convenience Score | 66.23 (21.451) | 66.02 (23.017)
  Overall Satisfaction Score | 64.23 (29.401) | 63.51 (27.603)

45. Secondary Outcome: Placebo-controlled Period: Migraine Specific Health Care Resource Utilization (HCRU) - Visits to a Family Doctor/General Practitioner at Baseline and Week 12
Description: Number of participants who visited to a family doctor/general practitioner during the past 4 weeks has been reported at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 288 | 281
Participants
  Baseline: number analyzed (Participants) | 283 | 267
  Baseline: 0 Visit | 213 | 198
  Baseline: 1 Visit | 44 | 42
  Baseline: 2 Visits | 10 | 17
  Baseline: 3 Visits | 11 | 4
  Baseline: 4 Visits | 2 | 3
  Baseline: 5 Visits | 1 | 2
  Baseline: 6 Visits | 1 | 0
  Baseline: 10 Visits | 1 | 0
  Baseline: 15 Visits | 0 | 1
  Week 12: 0 Visit | 242 | 217
  Week 12: 1 Visit | 29 | 41
  Week 12: 2 Visits | 7 | 15
  Week 12: 3 Visits | 5 | 4
  Week 12: 4 Visits | 4 | 2
  Week 12: 5 Visits | 0 | 2
  Week 12: 6 Visits | 1 | 0
  Week 12: 10 Visits | 0 | 0
  Week 12: 15 Visits | 0 | 0

46. Secondary Outcome: Placebo-controlled Period: Migraine Specific HCRU - Visits to a Specialist at Baseline and Week 12
Description: Number of participants who visited a specialist during the past 4 weeks has been reported at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 288 | 281
Participants
  Baseline: number analyzed (Participants) | 283 | 267
  Baseline: 0 Visit | 180 | 156
  Baseline: 1 Visit | 71 | 83
  Baseline: 2 Visits | 21 | 18
  Baseline: 3 Visits | 6 | 5
  Baseline: 4 Visits | 3 | 2
  Baseline: 5 Visits | 1 | 2
  Baseline: 6 Visits | 1 | 0
  Baseline: 12 Visits | 0 | 1
  Week 12: 0 Visit | 245 | 224
  Week 12: 1 Visit | 30 | 43
  Week 12: 2 Visits | 7 | 8
  Week 12: 3 Visits | 1 | 5
  Week 12: 4 Visits | 4 | 1
  Week 12: 5 Visits | 1 | 0
  Week 12: 6 Visits | 0 | 0
  Week 12: 12 Visits | 0 | 0

47. Secondary Outcome: Placebo-controlled Period: Migraine Specific HCRU - Number of Emergency Department Visits Due to Migraine at Baseline and Week 12
Description: Number of participants who visited to the emergency department due to migraine during the past 4 weeks has been reported at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 288 | 281
Participants
  Baseline: number analyzed (Participants) | 283 | 267
  Baseline: 0 Visit | 275 | 256
  Baseline: 1 Visit | 7 | 7
  Baseline: 2 Visits | 1 | 3
  Baseline: 9 Visits | 0 | 1
  Week 12: 0 Visit | 281 | 268
  Week 12: 1 Visit | 5 | 10
  Week 12: 2 Visits | 2 | 3
  Week 12: 9 Visits | 0 | 0

48. Secondary Outcome: Placebo-controlled Period: Migraine Specific HCRU - Number of Hospital Admissions Migraine at Baseline and Week 12
Description: Number of participants who were admitted to the hospital during the past 4 weeks due to migraine has been reported at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 288 | 281
Participants
  Baseline: number analyzed (Participants) | 283 | 267
  Baseline: 0 Admission | 279 | 258
  Baseline: 1 Admission | 3 | 7
  Baseline: 2 Admissions | 1 | 1
  Baseline: 16 Admissions | 0 | 1
  Week 12: 0 Admission | 286 | 277
  Week 12: 1 Admission | 2 | 4
  Week 12: 2 Admissions | 0 | 0
  Week 12: 16 Admissions | 0 | 0

49. Secondary Outcome: Placebo-controlled Period: Migraine Specific HCRU - Total Number of Participants With Overnight Hospital Stays Due to Migraine at Baseline and Week 12
Description: Number of participants who had overnight hospital stays during the past 4 weeks due to migraine has been reported at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo
Number analyzed (Participants) | 288 | 281
Participants
  Baseline: number analyzed (Participants) | 283 | 267
  Baseline: 0 Stay | 282 | 264
  Baseline: 1 Stay | 1 | 1
  Baseline: 2 Stays | 0 | 1
  Baseline: 7 Stays | 0 | 1
  Week 12: 0 Stay | 287 | 278
  Week 12: 1 Stay | 1 | 3
  Week 12: 2 Stays | 0 | 0
  Week 12: 7 Stays | 0 | 0

50. Secondary Outcome: Open-label Period: Migraine Specific HCRU - Visits to a Family Doctor/General Practitioner at Week 24
Description: Number of participants who visited a family doctor/general practitioner has been reported.
Time Frame: Week 24
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 281 | 275
Participants
  0 Visit | 239 | 239
  1 Visit | 26 | 20
  2 Visits | 11 | 13
  3 Visits | 3 | 1
  4 Visits | 1 | 0
  5 Visits | 0 | 1
  7 Visits | 0 | 1
  8 Visits | 0 | 0
  13 Visits | 1 | 0

51. Secondary Outcome: Open-label Period: Migraine Specific HCRU - Visits to a Specialist at Week 24
Description: Number of participants who visited a specialist has been reported.
Time Frame: Week 24
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 281 | 275
Participants
  0 Visit | 239 | 240
  1 Visit | 29 | 20
  2 Visits | 7 | 8
  3 Visits | 3 | 4
  4 Visits | 1 | 2
  5 Visits | 0 | 1
  6 Visits | 1 | 0
  7 Visits | 1 | 0

52. Secondary Outcome: Open-label Period: Migraine Specific HCRU - Number of Participants With Emergency Department Visits Due to Migraine at Week 24
Description: Number of participants who visited the emergency department due to migraine has been reported.
Time Frame: Week 24
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 281 | 275
Participants
  0 Visit | 277 | 265
  1 Visit | 3 | 5
  2 Visits | 0 | 3
  3 Visits | 0 | 1
  10 Visits | 0 | 1
  18 Visits | 1 | 0

53. Secondary Outcome: Open-label Period: Migraine Specific HCRU - Number of Participants With Hospital Admissions Due to Migraine at Week 24
Description: Number of participants who admitted in the hospital due to migraine has been reported.
Time Frame: Week 24
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 281 | 275
Participants
  0 Admission | 281 | 271
  1 Admission | 0 | 2
  2 Admissions | 0 | 2

54. Secondary Outcome: Open-label Period: Migraine Specific HCRU - Number of Participants With Overnight Hospital Stays Due to Migraine at Week 24
Description: Number of participants with overnight hospital stays due to migraine has been reported.
Time Frame: Week 24
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Period: Eptinezumab - Eptinezumab | Open-label Period: Placebo - Eptinezumab
Number analyzed (Participants) | 281 | 275
Participants
  0 Stay | 281 | 270
  1 Stays | 0 | 3
  2 Stays | 0 | 1
  12 Stays | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 32 weeks
Groups:
- Placebo-controlled Period: Placebo: Participants received an IV infusion of placebo at Baseline (Week 0) during the placebo-controlled period.
- Open-label Period: Eptinezumab to Eptinezumab; Open-label Period: Placebo to Eptinezumab: Participants who received eptinezumab during the placebo-controlled period received eptinezumab during the open-label period.
Arm/Group | Placebo-controlled Period: Eptinezumab | Placebo-controlled Period: Placebo | Open-label Period: Eptinezumab to Eptinezumab | Open-label Period: Placebo to Eptinezumab
All-Cause Mortality (participants affected / at risk) | 0/303 | 0/301 | 0/300 | 0/293
Serious Adverse Events (participants affected / at risk) | 2/303 | 1/301 | 2/300 | 5/293
Other Adverse Events (participants affected / at risk) | 50/303 | 55/301 | 30/300 | 42/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-controlled Period: Eptinezumab (N=303) | Placebo-controlled Period: Placebo (N=301) | Open-label Period: Eptinezumab to Eptinezumab (N=300) | Open-label Period: Placebo to Eptinezumab (N=293)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-controlled Period: Eptinezumab (N=303) | Placebo-controlled Period: Placebo (N=301) | Open-label Period: Eptinezumab to Eptinezumab (N=300) | Open-label Period: Placebo to Eptinezumab (N=293)
Asthenia (General disorders) | 3 (3) | 3 (3) | 1 (1) | 6 (6)
Fatigue (General disorders) | 6 (7) | 11 (11) | 6 (6) | 5 (6)
COVID-19 (Infections and infestations) | 6 (6) | 4 (4) | 5 (5) | 6 (6)
Influenza (Infections and infestations) | 11 (12) | 10 (10) | 7 (7) | 6 (7)
Nasopharyngitis (Infections and infestations) | 15 (16) | 17 (18) | 7 (8) | 10 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (8) | 3 (3) | 4 (4)
Dizziness (Nervous system disorders) | 8 (9) | 9 (12) | 1 (1) | 8 (10)
Insomnia (Psychiatric disorders) | 2 (2) | 8 (8) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT05452239/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT05452239/SAP_001.pdf